CLINICAL TRIAL: NCT05692765
Title: Effects of a Smartphone Application on Fruit and Vegetable Consumption Among Saudi Adolescents: A Randomized Intervention Study
Brief Title: Effects of a Smartphone Application on Fruit and Vegetable Consumption Among Saudi Adolescents
Acronym: F&V intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Israa Shatwan, Dr, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: reference number: 101-21
Record Dates: First submitted 2023-01-09; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Fruit and Vegetable Intake

STUDY DESIGN:
Intervention Model Description: This was a randomized intervention study conducted on 104 adolescents: 49 in the control group and 55 in the intervention group. The researcher provided a brief presentation about the health benefits and appropriate serving sizes of F&Vs and explained how to use the smartphone application. An instructional brochure was provided in Arabic to all adolescents in the intervention group. The participants in the intervention group were required to choose three of seven goals for each F&V.After choosing six goals (three for fruit and three for vegetables), the participants were required to mark the goal that they chose daily and were requested to adhere to their chosen goals until the end of the study. They were encouraged to turn on notifications for the application to receive reminder messages. Adolescents in the control group were not exposed to the smartphone application and did not receive any advice to promote their F&V consumption, which may have affected their F&V consumption.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Adolescents in the control group were not exposed to the smartphone application and did not receive any advice to promote their F&V consumption, which may have affected their F&V consumption. Instead, they were only asked to complete the pre- and post-questionnaires.
- Intervention group (Experimental): Adolescents in the intervention group were divided into 11 smaller groups, each containing five participants to explain the application. The researcher provided a brief presentation about the health benefits and appropriate serving sizes of F&Vs and explained how to use the smartphone application. An instructional brochure was provided in Arabic to all adolescents in the intervention group. The research team was available to assist participants at any time during the study period. After choosing six goals (three for fruit and three for vegetables), the participants were required to mark the goal that they chose daily and were requested to adhere to their chosen goals until the end of the study. The intervention period was 6 weeks.
  Interventions: Behavioral: smartphone application to enhance fruit and vegetables intake among adolescents

INTERVENTIONS:
Behavioral: smartphone application to enhance fruit and vegetables intake among adolescents — This randomized intervention study was conducted in an urban area of Jeddah, Saudi Arabia. We included 104 adolescents aged 13-18 years, who were randomized into intervention (n=55) or control (n=49) arms. We examined the effects of a smartphone application ("My Plate") on fruit and vegetable intake over 6 weeks in the intervention group. Pre- and postintervention questionnaires were used in the intervention and control groups.
  Arms: Intervention group

SUMMARY:
Background: Dietary patterns and nutritional status during adolescence have a direct effect on future health outcomes.

Objective: This study aimed to promote fruit and vegetable intake among adolescents using a smartphone application called "MyPlate." Methods: This randomized intervention study was conducted in an urban area of Jeddah, Saudi Arabia. The sample included 104 adolescents aged 13-18 years, who were randomized into intervention (n=55) or control (n=49) arms. The effects of a smartphone application ("My Plate") on fruit and vegetable intake was examined over 6 weeks in the intervention group. Pre- and postintervention questionnaires were used in the intervention and control groups.

DETAILED DESCRIPTION:
Participants and Recruitment This randomized intervention study was conducted between February and March 2021 among adolescents from Jeddah, Saudi Arabia. Since schools were closed because of the coronavirus disease 2019 pandemic, adolescents were recruited through invitations sent via emails and WhatsApp application to their parents using snowballing recruitment. The invitation to the study was first sent to members and Bachelor of Science students of the Food and Nutrition Department at King Abdulaziz University to help the research team with recruitment. Then, the research team contacted the parents and adolescents who voluntarily agreed to participate in the study. The study procedures were explained to the parents or guardians of all prospective participants. There were no imposed circulation restrictions or curfews in Jeddah during the study period. The inclusion criteria were healthy boys and girls (based on the self-reported absence of diseases, such as diabetes mellitus, that may influence food intake) aged 13-18 years, at schools, and able to use smartphones, either their own or their parents. The exclusion criteria were unhealthy adolescents or those not within the age range of this study. In total, 146 adolescents were initially recruited, of which 26 withdrew from the study because they did not complete the baseline questionnaire or voluntarily decided to withdraw. The remaining 120 adolescents were randomly divided into intervention and control groups. Microsoft Excel (version 22, Microsoft Corp., Redmond, WA, USA) with the RAND function was used to randomize the sample. After generating a random number, the participants were divided into control and intervention groups. As 16 adolescents decided not to complete the study or did not fill in the final questionnaire, 104 adolescents (24 boys and 80 girls) completed the intervention phase of the study.

The sample size was determined based on the ability to detect an expected mean difference of .7 servings according to a previous parallel intervention study [18] with 80% power and a 5% significance level. The calculated required sample size was 33 adolescents in each group [19]. Thus, considering a nearly 50% drop-out rate, we recruited 60 participants for each group. Study procedures were approved by the Unit of Biomedical Ethics Research Committee at King Abdulaziz University (reference number: 101-21). All adolescents were voluntarily recruited and provided verbal consent for participation in the study; their parents or guardians provided written informed consent.

Study Design This was a randomized intervention study conducted on 104 adolescents: 49 in the control group and 55 in the intervention group. Adolescents in the intervention group were divided into 11 smaller groups, each containing five participants to explain the application. One of the researchers conducted video conference calls with each of these small intervention groups. The researcher provided a brief presentation about the health benefits and appropriate serving sizes of F&Vs and explained how to use the smartphone application. An instructional brochure was provided in Arabic to all adolescents in the intervention group. The research team was available to assist participants at any time during the study period. The participants were required to choose three of seven goals for each F&V. The fruit goals were as follows: (1) have fruit with dinner; (2) add fruit to your salad; (3) snack on fruit; (4) have fruit for a sweet treat; (5) have fruit with lunch; (6) add frozen, canned, or dried fruit to your meal; and (7) start your day with fruit. The vegetable goals were as follows: (1) have vegetables with dinner; (2) have a dark green vegetable; (3) start your day with vegetables; (4) have a red or orange vegetable; (5) have vegetables with lunch; (6) snack on vegetables; and (7) make a salad or side dish using beans, peas, or lentils. After choosing six goals (three for fruit and three for vegetables), the participants were required to mark the goal that they chose daily and were requested to adhere to their chosen goals until the end of the study. They were encouraged to turn on notifications for the application to receive reminder messages. The research team also sent weekly WhatsApp text message reminders (in Arabic language) to the adolescents. The intervention period was 6 weeks. Adolescents in the control group were not exposed to the smartphone application and did not receive any advice to promote their F&V consumption, which may have affected their F&V consumption. Instead, they were only asked to complete the pre- and post-questionnaires.

This study used the free nutritional "MyPlate" smartphone application which is readily available on both iOS and Android platforms to promote F&V intake among adolescents. The application is a multi-component communications plan that was developed by the US Department of Agriculture Food and Nutrition Service in 2011. The app aids in translating the American Dietary Guidelines to the public and can be used as a nutritional education resource for children and adults. The application icon is an easy, effective, visual platform that helps promote healthy food choices, including all food groups, and create a balanced plate at mealtimes. The application allows one to set daily healthy eating goals for each food group and track individual progress [15,16]. Additionally, the Saudi dietary guidelines (including healthy Saudi plate) have been developed based on evidence from several dietary guidelines including the American dietary guidelines [20]. Since no Arabic applications are available in smartphone stores with similar features, we used the "MyPlate" application in the current study.

Data Collection All measures were collected via an online questionnaire on Google Forms. The questionnaire consisted of two parts. The first part included sociodemographic data, including information regarding age, sex, school type (private or public), weight and height of the adolescents and their parents, parents' education level (high school or lower, bachelor's degree, or postgraduate degree), parents' occupation (employed or unemployed), number of children in the family, and family income. This part of the questionnaire was completed by the participant with the assistance of one of their parents. The research team provided instructions to participants on the appropriate way to measure height and weight using a weight scale and measuring tape. Body mass index (BMI) was calculated as the weight in kilogram divided by the height in meters squared (kg/m2). BMI was evaluated using the Saudi growth chart (BMI-for-age). A BMI between the 15th and 85th percentile was considered normal; between the 85th and 95th percentile was considered overweight, and above the 95th percentile indicated obesity [21].

Fruit and Vegetable Consumption Questionnaires A validated food frequency questionnaire (FFQ) was used to compare F&V consumption in adolescents at baseline and after the intervention period in both groups. The FFQ was previously used with some adaptations to make it suitable for Saudi adolescents [13,18]. The response for each F&V item was recorded over seven frequency options (never, 1-3 times per month, 1 or 2 times per week, 3-4 times per week, 5-6 times per week, once per day, or 2 or more times per day). In total, 22 FFQ items were directly related to vegetable intake, whereas 18 FFQ items were directly related to fruit intake (Supplementary Table 1 shows the F&Vs listed in the FFQ). The response for each F&V item had seven frequency options; thus, it was scored based on a seven-scale grade. The highest score was 7 for two or more per day, and the lowest score was zero (never). The F&V scores were calculated separately, and the sum of the scores for all fruit items for each participant was divided by the total number of fruit items in the FFQ (18) and similarly for vegetable scores.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were healthy boys and girls (based on the self-reported absence of diseases, such as diabetes mellitus, that may influence food intake) aged 13-18 years, at schools, and able to use smartphones, either their own or their parents.

Exclusion Criteria:

* The exclusion criteria were unhealthy adolescents or those not within the age range of this study.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetables intake | 6 weeks
  measuring score difference of fruit and vegetables consumption before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Food and Nutrition department, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shatwan IM, Alhefani RS, Bukhari MF, Hanbazazah DA, Srour JK, Surendran S, Aljefree NM, Almoraie NM. Effects of a Smartphone App on Fruit and Vegetable Consumption Among Saudi Adolescents: Randomized Controlled Trial. JMIR Pediatr Parent. 2023 Feb 9;6:e43160. doi: 10.2196/43160. PMID 36757770